CLINICAL TRIAL: NCT04312529
Title: Analysis of Shoulder Muscle Activity During Isokinetic Evaluation of Rotators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Principal investigator, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1996
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Muscle Activation; Electromyography; Muscle Strength; Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overhead athletes (Experimental)
  Interventions: Other: Isokinetic test + EMG

INTERVENTIONS:
Other: Isokinetic test + EMG — Isokinetic test:The isokinetic device is used to evaluate the strength of a subject. The test will be performed in two positions. This will determine the best position to activate shoulder muscles EMG (electromyography):it's a device that measures the electrical activity of muscles. This will allow us to record the maximum activity of the shoulder muscles during force tests.

SUMMARY:
The objective of this study is to assess the impact of different positions of the glenohumeral joint on the maximum muscle contraction of different shoulder muscles. The muscles do not contract with the same intensity depending on the position of the arm in relation to the trunk. With the determination of this optimal position to activate the shoulder muscles as much as possible, we will be able to strengthen the patients during their revalidation.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-35.
* Playing a sport using the upper limb (handball, volleyball, swimming, tennis) at least 6h/week

Exclusion Criteria:

* Pain in the shoulder
* Shoulder pathologies such as gleno-humeral dislocation, tendinopathy, sub-acromial conflict, etc.
* History of shoulder surgery (prosthesis, stabilizing surgery, etc.)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
strength test | Day 1.
  The strength will be assess with a isokinetic device. It will allow to calculate the maximum force of the subject at the level of the rotators of the shoulder. This is a dorsal decubitus test. The subject's arm will be positioned during one session in 45° of abduction and the other session in 90° of shoulder abduction.
  In this position, the subject will perform tests at different speeds (60°/s concentric, 240°/s concentric and 60°/s eccentric). This will calculate the maximum force.
Electrical activity of the muscles | Day 1.
  The electromyography will allow to calculate the electrical activity of the muscles during the two isokinetics and thus to determine which active position the most the muscles of the shoulder. This measurement is achieved by the installation of surface electrodes

SECONDARY OUTCOMES:
Weight | Day 1
  We will ask the weight of the subject to calculate his relative strength

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Liège, Liège, Belgium